CLINICAL TRIAL: NCT02471950
Title: The Depth of Anaesthesia Associated With the Use of 2.5% Isoflurane During Cardiopulmonary Bypass
Brief Title: Isoflurane During Cardiopulmonary Bypass
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 15 LO 0366; 2015/0199 (Other: NHS Lothian)
Record Dates: First submitted 2015-06-01; First posted 2015-06-15 (Estimated); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Cardiopulmonary Bypass; Consciousness Monitors; Isoflurane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Arterial and venous blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Elective Cardiac surgery: Those patients scheduled for elective heart surgery requiring cardiopulmonary bypass who will be given 2.5% isoflurane while on bypass.
  Interventions: Procedure: 2.5 % Isoflurane administration

INTERVENTIONS:
Procedure: 2.5 % Isoflurane administration — Anaesthesia maintained during cardiopulmonary bypass with 2.5% isoflurane administered via the oxygenator of the bypass circuit.

SUMMARY:
There is no clinical way of assessing the depth of anaesthesia while patients are on the heart-lung machine. A new method of measuring the depth of anaesthesia using brainwaves called the Bispectral index (BIS) has been developed and its use in cardiac surgery is now widespread. However BIS is also altered by patients body temperature. As cooling is common during heart surgery the use of BIS to measure the depth of anaesthesia during heart-lung bypass remains controversial. This study aims to find out what depth of anaesthesia is produced according to BIS during heart lung bypass using a standard anaesthetic technique that utilises the anaesthetic isoflurane.

DETAILED DESCRIPTION:
There is no clinical way of assessing patients' depth of anaesthesia on the heart-lung machine. For this reason, the amount of volatile anaesthetic agent like isoflurane, that is administered has traditionally been determined by anaesthetists' clinical experience. Recently, a device that assesses depth of anaesthesia by analysing the electrical brain waves called the Bispectral index (BIS) has been introduced. The study aims to determine whether the level of anaesthesia produced by isoflurane using the traditional approach is more than required simply to maintain unconsciousness according to BIS. In addition, the study will determine whether the concentration of isoflurane in exhaust gases from the heart-lung machine can be used as an estimate arterial blood concentration and so, depth of anaesthesia.

The study will recruit patients who are scheduled for heart surgery using a heart-lung machine. Patients will be anaesthetised using a long established balanced technique including the administration of isoflurane 2.5% whilst supported on the heart-lung machine. Measurements of exhaust gas concentration of isoflurane from the heart-lung machine and level of BIS will be recorded at three time points. Simultaneously, three arterial blood samples will be taken and the isoflurane concentration measured in these samples. The BIS levels will be averaged and the proportion of patients with a BIS below 40 (lower limit of normal) will be calculated. Concentrations of isoflurane in the exhaust gas of the heart-lung machine will be compared with blood concentrations of isoflurane and the both concentrations will be compared with the level of BIS to establish whether they can be used to assess depth of anaesthesia.

If this study finds that a large proportion of patients have more than adequate levels of anaesthesia, then future studies could explore whether administering lower concentrations of isoflurane improves outcome whilst maintaining anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Participants over the age of 18
* Scheduled for elective cardiac surgery under the care of trial anaesthetists
* Patient has provided informed consent to participate

Exclusion Criteria:

* Patients presenting for emergency cardiac surgery
* Patients who will have cardiac surgery that does not require cardiopulmonary bypass
* Unwilling/unable to provide informed consent
* Patients under the age of 18
* Anaesthesia undertaken by anaesthetists not involved in trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those patients scheduled for elective heart surgery over the age of 18 requiring cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Depth of anesthesia according to BIS | Intraoperative
  BIS reading will be recorded at three time points during cardiopulmonary bypass

SECONDARY OUTCOMES:
Comparison of exhaust gas and blood concentration of isoflurane | Intraoperative
  Exhaust gas and blood concentrations of isoflurane will be recorded at three time points during the operation. These values will be compared to see if their values are are related.
Comparison of blood isoflurane concentration and BIS score | Intraoperative
  Blood isoflurane concentration and BIS will be recorded at three time points and compared to see if they are related
Comparison of exhaust isoflurane Concentration and BIS score | Intraoperative
  Exhaust isoflurane and BIS will be recorded at three time points and compared to see they are related.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Alston, MBChB, Principal Investigator — University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Scotland, United Kingdom

REFERENCES:
- [Result] Alston RP, Connelly M, MacKenzie C, Just G, Homer N. The depth of anaesthesia associated with the administration of isoflurane 2.5% during cardiopulmonary bypass. Perfusion. 2019 Jul;34(5):392-398. doi: 10.1177/0267659118822946. Epub 2019 Jan 12. PMID 30638148